CLINICAL TRIAL: NCT03382314
Title: A Randomized, Open-label, Single-dose, Crossover Study to Evaluate the Pharmacokinetic Characteristics After Co-administration of HDDO-16141 and HDDO-16143 and Administration of HDDO-1614 in Healthy Adult Male Subjects
Brief Title: HDDO-1614 Bio Equivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hyundai Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HT-008-02
Record Dates: First submitted 2017-12-07; First posted 2017-12-22 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — bazedoxifene; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HDDO-1614 (Experimental): Bazedoxifene + Cholecalciferol combination drug
  Interventions: Combination Product: HDDO-1614
- Bazedoxifene + Cholecalciferol (Active Comparator): Co-administration of Bazedoxifene and Cholecalciferol
  Interventions: Drug: Bazedoxifene / Cholecalciferol

INTERVENTIONS:
Combination Product: HDDO-1614 — * Combination drug (Bazedoxifene + Cholecalciferol)
  * Incrementally modified drug
  * Not market authorized product
  Arms: HDDO-1614
Drug: Bazedoxifene / Cholecalciferol — Co- Administration of Bazedoxifene and Cholecalciferol
  Arms: Bazedoxifene + Cholecalciferol

SUMMARY:
A randomized, open-label, single-dose, crossover study

DETAILED DESCRIPTION:
This clinical trial is conducted with a randomized, open-label, single-dose, and cross over study designs. Investigators will compare the pharmacokinetic parameters of test drug(single oral dose, single administration) with pharmacokinetic parameters of comparator 1 and 2(combined administration, single oral dose).

ELIGIBILITY:
Inclusion Criteria:

* Body weight 50kg ≤ / BMI=18~29kg/㎡
* A person who is determined to be eligible for the test through a physical examination or an interview
* Those who have been judged to be eligible for the clinical laboratory tests such as hematology test, blood chemistry test, urine test, and serology test

Exclusion Criteria:

* Patients with clinically significant liver, pancreas, kidney, nervous system, respiratory, endocrine, hematologic, mental, cardiovascular
* Patients with a history of gastrointestinal disorders or history of gastrointestinal surgery that may affect the absorption of pharmaceuticals for clinical trials
* Any person who shows any of the following results in the screening test

  1. AST or ALT > 2 times upper limit of normal range
  2. Total Bilirubin > 2.0mg/dL
  3. Glomerular filtration Rate(eGFR) < 60mL/min/1.7㎡
* Those who show signs of hypotension (systolic blood pressure ≤ 100mm Hg or diastolic blood pressure ≤ 55mmHg) or Hypertension (systolic blood pressure ≥ 150mmHg or diastolic blood pressure ≥ 95mmHg)
* Those who have a history of drug or who have a positive urine drug test

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2018-01-05 (Actual)

PRIMARY OUTCOMES:
Bio-Equivalence between test drug and comparators | Day 1 ~ Day 27
  To evaluate the bio-equivalence between co-administration of Bazedoxifene and Cholecalciferol and administration of HDDO-1614

SECONDARY OUTCOMES:
Bazedoxifene Pharmacokinetic Assessment | 0, 0.333, 0.667, 1, 1.5, 2, 3, 4, 6, 12, 24, 48, 72, 96 and 120 hours
  Bazedoxifene Maximum Plasma Concentration
Cholecalciferol Pharmacokinetic Assessment | Pre-dose: -24, -18, -12, 0 hour, Post-dose: 2, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48, 72, 96 hour
  Maximum Plasma Concentration after correction of basal concentration of Cholecalciferol

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Junggu, Incheon, South Korea